CLINICAL TRIAL: NCT03931135
Title: Comparison Between Cyclizine and Dexamethasone for Prevention of Nausea and Vomiting After Intrathecal Morphine in Patients Undergoing Cesarean Section
Brief Title: Cyclizine Vs. Dexamethasone for Nausea and Vomiting Following Intrathecal Morphine in Cases of Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Elia Azmy Habib, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cyclizine vs dexa for PONV
Record Dates: First submitted 2019-03-26; First posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-03

CONDITIONS: Spinal Anesthetics Causing Adverse Effects in Therapeutic Use

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Active Comparator)
  Interventions: Drug: IV Cyclizine versus IV Dexamethasone for prevention of nausea and vomiting after intrathecal morphine in patients undergoing cesarean section
- Cyclizine (Active Comparator)
  Interventions: Drug: IV Cyclizine versus IV Dexamethasone for prevention of nausea and vomiting after intrathecal morphine in patients undergoing cesarean section

INTERVENTIONS:
Drug: IV Cyclizine versus IV Dexamethasone for prevention of nausea and vomiting after intrathecal morphine in patients undergoing cesarean section — The first group (Dexamethasone) will receive 8 mg IV dexamethasone within 1-2 minutes after the umbilical cord is clamped.
  The second group (Cyclizine) will receive 50 mg cyclizine within 1-2 minutes after the umbilical cord is clamped

SUMMARY:
Comparing between cyclizine and dexamethasone in preventing PONV after CS under spinal anesthesia with spinal opiate.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is defined as any nausea, retching, or vomiting occurring during the first 24-48 h after surgery in patients. PONV is one of the most common causes of patient dissatisfaction after anesthesia, with reported incidences of 30% in all post-surgical patients and up to 80% in high-risk patients. In addition, PONV is regularly rated in preoperative surveys, as the anesthesia outcome the patient would most like to avoid. While suture dehiscence, aspiration of gastric contents, esophageal rupture, and other serious complications associated with PONV are rare, nausea and vomiting is still an unpleasant and all-too-common postoperative morbidity that can delay patient discharge from the post-anesthesia care unit and increase unanticipated hospital admissions in outpatients.

There are many well-established risk factors for PONV which are classified in two classes:

A) Patient related risk factors:

1. Female gender is consistently the strongest risk factor for PONV, female patient are three times more likely than men to suffer from PONV.
2. For adult patient, age is a statistically, though not clinically, relevant risk factor, with the incidence of PONV decreasing as patients age. For pediatric patients, however, age increases the risk of post-operative vomiting (POV), such that children older than 3 years have been shown to have an increased risk of POV compared with children younger than 3 years.
3. Obesity is a strong risk factor for PONV: patients with body mass index (BMI) more than 30 have the double risk of PONV.
4. Non-smoking status roughly doubles the patient's risk of PONV. The specific mechanism underlying smoking's protective effect is unknown ,but one of the most commonly believed theories is that polycyclic aromatic hydrocarbons in cigarette smoke induce cytochrome P450 enzyme which increase the metabolism of emetogenic volatile anesthetics.
5. History of gastrointestinal disease as gastritis, gastric ulcer or duodenal ulcer increases the risk for PONV.
6. History of motion sickness, Meniere's disease or previous PONV indicates a general susceptibility to PONV.

B) Anesthesia related risk factors:

1. The use of volatile anesthetics is associated with a two-fold increase in the risk of PONV, with risk increasing in a dose dependent manner.
2. Intraoperative and postoperative opioid use increases the risk of PONV in a dose dependent manner by the mechanism of reducing muscle tone and peristaltic activity, thereby delaying gastric emptying, inducing distention, and triggering the vomiting reflex.
3. The duration of anesthesia can help predict the patient's risk of PONV, since the duration of anesthesia describes the patient's exposure to emetogenic stimuli like volatile anesthetics and intraoperative opioids.

Anti-emetic drugs used to treat PONV:

1. The first line is classified into three classes: serotonin antagonists (e.g. ondansetron), corticosteroids (e.g. dexamethasone), and dopamine antagonists (e.g. droperidol) have similar efficacy against PONV, with a relative risk reduction of about 25%. Moreover, they act independently and when used in combination, have additiveeffects.

   Dexamethasone : it can be effective in preventing PONV in adults and children. Compared with other operative medications, dexamethasone has equal or even better efficacy in reducing the incidence of PONV and has the advantages of low cost and longer effectiveness as well. The mechanism of the antiemetic action of dexamethasone is still not clearly known. Glucocorticoids receptors are found in nucleus of the solitary tract, the raphe nucleus and the area postrema and all are associated with regulating nausea and vomiting. Dexamethasone may affect PONV by modulating neurotransmission or receptor density in these nuclei. Clinically, dexamethasone as a preventive drug against PONV has not caused fatal outcome; therefore, it is generally considered to be an effective and safe anti-emetic. Nevertheless, its use in this regard may lead to adverse effects, principally postoperative hyperglycemia and infection.
2. The second line is Cyclizine: a histamine H1 antagonist given by mouth or parenterally for control of postoperative and drug-induced nausea and vomiting and in motion sickness. additionally, it has been used in management of vertigo in diseases affecting the vestibular apparatus. Although the mechanism by which cyclizine exerts its antiemetic and antivertigo effects has not been fully elucidated, its central anticholinergic properties are partially responsible. It also possesses anticholinergic, antihistaminic, central nervous system depressant and local anesthetic effects. cyclizine is metabolized to its N-demethylated derivative , norcyclizine , which has little antihistaminic activity compared to cyclizine.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 to 45 years old
* Parturient
* ASA I-II
* Full Term

Exclusion Criteria:

* Women who has obstetric complications.
* Women with evidence of foetal compromise.
* Patients who have gastro-intestinal diseases.
* Administration of anti-emetic drugs within 24 hours before operation.
* Patients who have hyperemesis gravidarium

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 160 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Post operative nausea and vomiting after intrathecal morphine by using PONV intensity scale. | Change in severity of nausea and vomiting 30 minutes , 3 hours, 6 hours after intervention
  Nausea and vomiting were recorded as present or absent,
  All measurements and ratings were completed at the time when patients rated their PONV intensity.
  We also recorded factors known to be associated with the risk of developing PONV, including known risk factors for PONV.

SECONDARY OUTCOMES:
Change in postoperative pain (assessed by VAS ). | Immediatly before and after intervention, 30 minutes after intervention, 3 hours after intervention, 6 hours
  0 meaning no pain at all, and 10 described as the worst pain experienced.

IPD SHARING:
Plan to Share IPD: Undecided